CLINICAL TRIAL: NCT03860649
Title: Effects of Different Physical Therapies and Dance on Clinical and Functional Parameters, Muscle Quality, Pendular Mechanism of the Gait and Brain-derived Neurotrophic Factor in People With Parkinson's Disease
Brief Title: Effects of Different Physical Therapies and Dance in People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Aline Nogueira Haas (Unknown); Flávia Gomes Martinez (Unknown)
Responsible Party: Principal Investigator, Leonardo A. Peyré-Tartaruga, Adjunct Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTartaruga,PPT-Parkinson
Record Dates: First submitted 2018-12-05; First posted 2019-03-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Parkinson Disease 10
Keywords: Mobility; Functionality; Movement disorders; Rehabilitation; Locomotion
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 10; Movement Disorders | interventions — Nordic Walking; Jogging; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: double-blind (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nordic Walking (Experimental): The patient walk program consists of 3 moments: warm up, walk and stretch. They will do a brief free walking warm-up for 3 minutes in the Self-selected walking speed - SSWS (3 'SSWS), then walk according to the training cycle, the intensity will be between 60 to 80% of the Heart of Ratio reserve. In addition, the intensity of the classes will be measured in each phase by the Borg Scale of Perceived Exertion.
  Interventions: Other: Nordic Walking
- Jogging (Experimental): This group will undergo 24 Dance sessions. Aquatic therapy patients will receive deep water running intervention with the use of flotation vests. The exercises will consist of: immersion, balance, strength, agility, and movement within the water. The intensity of the classes will be measured in each moment and by the Borg Scale of Perceived Exertion.
  Interventions: Other: Jogging
- Dance (Experimental): This group will undergo 24 Dance sessions inspired by Forró dance rhythm and Samba dance rhythm. Classes will be divided into four stages: Joint warm up and stretching on the chairs; strengthening, balance and rhythm exercises with the support of the barre; exercises inspired by the Samba and Forró dance (Brazilian ballroom dance) basic steps; and Final cool down. The intensity of the classes will be measured according to the beats per minute (BPMs) of the songs used in each moment and by the Borg Scale of Perceived Exertion.
  Interventions: Other: Dance
- Pilates Training (Experimental): Classes composed of three phases: Warming up, main part and back to calm. Warming up will begin with pre-Pilates training exercises for 5 minutes (eg. breathing exercises, hip joint mobilization, shoulder girdle, etc.), the main part of the lesson will be the Pilates training drill sequence for the beginner level that will be conducted for 50 minutes in which all exercises will be performed on the floor.
  The sequence of the eighteen exercises of the main part of the lesson is described in the table below. Back to Calm: will be carried out for 5 final minutes with standing exercises with the subject reclining on the wall to reconnect the subject with orthostatic posture.
  In the each of the phases of the lesson will be shown to the subject the table of BORG with the objective of measuring the intensity of perceived exertion, using the Borg Scale of Perceived Exertion.
  Interventions: Other: Pilates Training

INTERVENTIONS:
Other: Nordic Walking — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Nordic Walking
Other: Jogging — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Jogging
Other: Dance — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Dance
Other: Pilates Training — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Pilates Training

SUMMARY:
The aim of study is to analyze the effects of different physical therapies (Aquatic Jogging, Neurofunctional Physiotherapy, Pilates Training and Nordic Walking) and Dance and compare with unsupervised home exercises in the clinical-functional parameters, postural balance, muscular echographic quality, pendulum gait mechanism, and serum levels of BDNF in people with Parkinson's disease with camptocormia or Pisa Syndrome.

DETAILED DESCRIPTION:
Objective: Analyze the effects of different physical therapies (Aquatic Jogging, Neurofunctional Physiotherapy, Pilates Training and Nordic Walking) and Dance and compare with unsupervised home exercises in the clinical-functional parameters, postural balance, muscular echographic quality, pendulum gait mechanism, and serum levels of brain-derived neurotrophic factor (BDNF) in people with Parkinson's disease with camptocormia or Pisa Syndrome. Experimental Design: Randomized controlled clinical trial with translational study characteristics. Search Location: Exercise Research Laboratory at the School of Physical Education, Physiotherapy and Dance, Federal University of Rio Grande do Sul, and in the Movement Disorders Outpatient Clinic of the Hospital of Clinicals of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil. Participants: 100 patients from the Unified Health System (UHS) of both sexes, from 50 to 80 years old, diagnosed with idiopathic PD, sedentary. Interventions: In this research, four groups of patients with PD will receive intervention during 4 months of different physical therapy programs (Nordic walking, aquatic jogging and supervised neurofunctional physiotherapy) and dance; and a control group, who will receive telephone guidance for performing home-based exercises. The training programs will have a duration of 4 months and will be periodized so that the duration of the sessions is matched between them. The intensity of the interval training will be manipulated by the subjective effort scale (Borg) and by the heart rate, with predetermined series durations. All training programs will have a frequency of two sessions per week and a duration of 60 minutes. In order to evaluate the effects of the training, evaluations will be performed before and after the training period: 1) Basal (month 0): initial pre-training evaluation; 2) month 4: Evaluation 48h after the last training session. Outcomes: clinical-functional parameters, postural balance, muscular echographic quality, pendulum gait mechanism, and biochemistry. Data Analysis: Data will be described by average values and standard deviation values. The comparisons between and within groups will be performed using a Generalized Estimating Equations (GEE) analysis, adopting a level of significance (α) of 0.05. Expected Results: The intervention groups of the different physical therapies and dance are expected to be more effective in all outcomes analyzed, especially improving functional mobility when compared to the control group of unsupervised home exercises. In addition, it is expected that the results of the research will be expandable and the possibility of future developments in the scientific, technological, economic, social and environmental fields and that they will be implemented in the Unified Health System (UHS).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* aged over 40 years
* both sexes
* clinical diagnosis of idiopathic PD
* PD staging between 1 and 4 in Hoehn and Yahr Scale (H&Y).

Exclusion Criteria:

* performing recent surgeries, deep brain stimulation (DBS - Deep Brain Stimulations);
* severe heart diseases, uncontrolled hypertension, myocardial infarction within a period of less than one year, being a pacemaker;
* stroke or other associated neurological diseases; insanity;
* prostheses in the lower limbs;
* without ambulation conditions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Test Timed Up and Go | Change from baseline at 12 weeks.
  Test Timed Up and Go This teste evaluate the mobility functional in three meters of self-selected speed (TUGSS) or at forced speed (TUGFS).

SECONDARY OUTCOMES:
Locomotor Rehabilitation Index | Change from baseline at 12 weeks.
  The Locomotor Rehabilitation Index (LRI) is a method of determining how close is the self-selected walking speed compared to the Optimum Speed. The results is given in %, and when LRI value is closer to 100 %, it indicates that the participants are closer to their theoretical optimal walking speed.
Self-selected walking speed | Change from baseline at 12 weeks.
  SSWS This outcome will be measure in test of walking treadmill.
Optimal Walking Speed (OPT) | Change from baseline at 12 weeks.
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill.
Quality of life (QoL): PDQ-39 | Change from baseline at 12 weeks.
  The quality of life will be measured by the Parkinson's Disease Questionnaire, with 39 questions (PDQ-39). PDQ-39 is a PD specific health status questionnaire comprising 39 items. Respondents are requested to affirm one of five ordered response categories according to how often, due to their PD, they have experienced the problem defined by each item. The total scores are ranging between 0 and 100 points, that a lower score represents a greater perception of quality of life.
Cognitive function - Montreal Cognitive Assessment | Change from baseline at 12 weeks.
  Montreal Cognitive Assessment (MoCA) is a brief screening tool for mild cognitive impairment. This evaluation accesses different cognitive domains and investigates the individual's abilities in the following areas: attention and concentration, executive functions, memory, language, visuoconstructive skills, conceptualization, calculation and orientation. The total score of the MoCA is 30 points, with a score of 26, or more, considered normal and less than 26 is considered cognitive impairment.
Cognitive function - Mini Mental State Examination | Change from baseline at 12 weeks.
  Mini-Mental State Examination (MMSE) is a screening tool, used to identify dementia, which provides information on different cognitive parameters, containing questions grouped into seven categories that assess specific cognitive functions: temporal orientation, spatial orientation, three word registration, attention and calculation, recall of three words, language and visual constructive ability. The MMSE score can range from zero to 30 points, in which a lower score indicates a higher degree of cognitive impairment.
Depressive symptoms | Change from baseline at 12 weeks.
  This outcome will be measure for the Geriatric Depression Scale - 15 item. The scale consists of 15 dichotomous questions in which participants are asked to answer yes or no in reference to how they felt over the past week (for instance, "Do the pacient feel that their life is empty?," Do the patient feel that their situation is hopeless?). Scores range from 0 to 15 with higher scores indicating more depressive symptoms.

OTHER OUTCOMES:
Motor symptoms | Change from baseline at 12 weeks.
  This outcome will be evaluated using Unified Parkinson's Disease Rating Scale (UPDRS). This Scale the clinician-scored monitored motor evaluation. Will be to considered 30% improvement in motor symptoms has been applied to identify "responsive people". The score in each item ranges from 0 to 4, and the indicates greater impairment by the disease and the minimum, normality. The 14 items in the motor vehicle (the numbering of which goes from 18 to 31).
Freezing of Gait | Change from baseline at 12 weeks.
  The freezing of gait questionnaire (FOG-Q) has 6 questions and a total score of 0 to 24. A higher score corresponds to the more severe presence of freezing of gait and a lower score is equivalent to a lower presence or absence of freezing of gait .
Balance Static | Change from baseline at 12 weeks.
  The force platform will be used for the anteroposterior displacement of the center of pressure (COP)- COPx (in centimeters) and mediolateral - COPy (in centimeters) of the pressure center.
Spatial Parameter - Stride length | Change from baseline at 12 weeks.
  This outcome is measure by stride length in meters. This parameter will be measure before and after the nordic walking, dance and jogging aquatic interventions.
Temporal Parameter - Swing time, contact time, time of balance | Change from baseline at 12 weeks.
  Swing time in seconds, contact time in seconds, time of balance in seconds. The percentage of contact time will be calculated to measure the duty factor in percentual.
  The swing and contact time in seconds will be aggregated to distance in meters to arrive at frequency (in Hetz). These parameters will be measure before and after the nordic walking, dance and jogging aquatic interventions.
Anthropometric data - Body mass | Change from baseline at 12 weeks.
  Body mass will be measure in kilograms before and after the nordic walking, dance and jogging aquatic interventions.
  These data will be measured in scale, stadiometer and anthropometric tape. All this parameters will be measure before and after the nordic walking, dance and jogging aquatic interventions.
Anthropometric data - Height | Change from baseline at 12 weeks.
  Height will be measure in meters before and after the nordic walking, dance and jogging aquatic interventions.
Anthropometric data - Circumference | Change from baseline at 12 weeks.
  Circumference of body will be measure in centimeters before and after the nordic walking, dance and jogging aquatic interventions.
Anthropometric data - Body Mass Index | Change from baseline at 12 weeks.
  Weight and height will be combined to report the body mass index in kg/m2. This parameter will be measure before and after the nordic walking, dance and jogging aquatic interventions.
Electromyographic Parameters | Change from baseline at 12 weeks.
  This outcome is measure is a composite for: mean amplitude, onset, offset and time of the signal and co-contraction of the muscles: vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) all variables in percentage. This outcome will be measured through measuring the electromyographic activation during treadmill walking tests using an electromyograph.
Parameters of Pendular Mechanism - Internal Work | Change from baseline at 12 weeks.
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The internal work is the mechanical energy fluctuations of the movement of limbs relative to the center of body mass (Wint, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Parameters of Pendular Mechanism: external work | Change from baseline at 12 weeks.
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The external work is energy fluctuations of the center of body mass with respect to the external environment or surroundings (Wext, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Parameters of Pendular Mechanism: total mechanical work | Change from baseline at 12 weeks.
  The transduction between the potential and kinetic mechanical energies of the center of body mass (called the "inverted pendulum" mechanism). The total mechanical work (Wtot =Wext + Wint) produced by a body during activity. These outcomes are measured by composite for:(external, internal mechanical work, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Parameters of Pendular Mechanism: Recovery | Change from baseline at 12 weeks.
  The mechanical energy exchange of the center of mass is quantified by the calculation of the percentage of reconversion of mechanical energy, called Recovery (R), which counts the form that the mechanical energy is saved through the pendulum mechanism of the locomotion. This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
Motor behavior by electromyographic activity | Change from baseline at 12 weeks.
  During the gait initiation, sit-to-stand movement and go up and down one step, the investigators will evaluate the anticipatory postural adjustments and compensatory postural adjustments. The electromyograph will be used to obtain electromyographic activity data of the spinal erector muscles, internal oblique, gluteus medius, rectus femoris, femoral biceps, medial gastrocnemius and tibialis anterior (in mV).
  All these parameters will be measured before and after Nordic walking, dance and jogging interventions.
Muscular activation | Change from baseline at 12 weeks.
  Muscular activation during phases of the gait cycle of people with Parkinson's disease through the electromyographic evaluation of the muscles of the spinal erector, internal oblique, gluteus medius, rectus femoris, femoral biceps, anterior tibialis and medial gastrocnemius during treadmill running. All participants will walk on a treadmill at selected walking speed. To identify electromyographic activity during the different gait cycles, the electromyograph will be synchronized with VICON (Vicon Motion Capture System - Oxford - USA, 1984).
Scapular and pelvis coordination parameters | Change from baseline at 12 weeks.
  The scapular girdle movement in angles will be measure, pelvic girdle in angles will be measure.
  The scapular girdle movement in angles will be aggregated to pelvic girdle in angles to arrive at continuous and discrete phases coordinations in angles.
  All these parameters will be measure before and after the nordic walking, dance and jogging aquatic interventions.
Angular variables | Change from baseline at 12 weeks.
  Tilt pelvic in angle, flexion and extension of trunk in angle, flexion and extension of hip in angle, flexion and extension of knee in angle, flexion and extension of ankle in angle, flexion and extension of shoulder in angle, abduction of shoulder in angle, flexion and extension of elbow in angle. All these angles variables will be measure in right and left limbs.
  Flexion and extension of shoulder in angle, abduction of shoulder in angle will be aggregated to flexion and extension of elbow in angle to arrive at asymmetry of upper limbs in angles.
  * Maximum flexion and extension angles of trunk, hip, knee, ankle, shoulder and elbow;
  * Maximum and minimum abduction of shoulder.
  * Range of motion of the trunk (in the sagittal plane) and pelvic and scapular (in the transverse plane) girdle.
Body Composition - Bone mineral density. | Change from baseline at 12 weeks.
  The body composition of the patient will be analyzed using the dual-energy X-ray absorptiometry (DEXA - Lunar Prodigy GE model Medical System, Milwaukee, WI, USA).
  The patient will be lying down in the 10 to 12 minutes until the test is complete. To prevent the movement of the lower limbs during passage of the reading rod of the velcro around the ankles and thighs. The patient can wear normal clothes as long as they have no metal charges or attachments.
Psychological parameters - Profile of Mood State | Change from baseline at 12 weeks.
  Profile of Mood States: This variable will be measure by the Brunel Mood Scale (BRUMS) that was developed to provide a quick assessment of mood states adult populations. The BRUMS has been demonstrated to have Cronbach alpha values above 0.70 and is a reliable tool used to measure the mood of Brazilian athletes. The instrument consisted of 24 items and six subscales assessing mood: tension, depression, anger, vigor, fatigue and confusion. Each item was rated on a Likert scale ranging from nothing (0) to extremely (4), where the respondent indicated how they were feeling at that moment. The results were calculated using the mean of the items in each subscale.
Quality of sleep - The Pittsburgh Sleep Quality Index | Change from baseline at 12 weeks.
  The Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 24 questions or items to be rated (0-3 for 20 items while 4 items are open-ended), 19 of which are self-reported and 5 of which require secondary feedback from a room or bed partner. Only the self-reported items (15 rated as 0-3 while 4 open-ended) are used for quantitative evaluation of sleep quality as perceived by the patient. The open-ended items are also finally scored as structured categorical values (rated at 0-3) as per the range of values reported for them by the patient. These 19 self-reported items are used to generate categorical scores representing the PSQI's 7 components. The individual component scores each assess a specific feature of sleep. Finally, the scores for each component are summed to get a total score, also termed the global score (range: 0 to 21). This score provides a summary of the respondent's sleep experience and quality for the past month.
Nominal verbal fluency | Change from baseline at 12 weeks.
  Nominal verbal fluency evaluates verbal fluency, executive function, language, and semantic memory. The test consists in naming the largest number of words beginning with the letters "F", "A" and "S" in one minute each, excluding proper names.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Alexandre Peyré-Tartaruga, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberts JL, Linder SM, Penko AL, Lowe MJ, Phillips M. It is not about the bike, it is about the pedaling: forced exercise and Parkinson's disease. Exerc Sport Sci Rev. 2011 Oct;39(4):177-86. doi: 10.1097/JES.0b013e31822cc71a. PMID 21799425
- [Background] Cavagna GA, Willems PA, Legramandi MA, Heglund NC. Pendular energy transduction within the step in human walking. J Exp Biol. 2002 Nov;205(Pt 21):3413-22. doi: 10.1242/jeb.205.21.3413. PMID 12324550
- [Background] Cho C, Kunin M, Kudo K, Osaki Y, Olanow CW, Cohen B, Raphan T. Frequency-velocity mismatch: a fundamental abnormality in parkinsonian gait. J Neurophysiol. 2010 Mar;103(3):1478-89. doi: 10.1152/jn.00664.2009. Epub 2009 Dec 30. PMID 20042701
- [Background] Dereli EE, Yaliman A. Comparison of the effects of a physiotherapist-supervised exercise programme and a self-supervised exercise programme on quality of life in patients with Parkinson's disease. Clin Rehabil. 2010 Apr;24(4):352-62. doi: 10.1177/0269215509358933. PMID 20360152
- [Background] Detrembleur C, van den Hecke A, Dierick F. Motion of the body centre of gravity as a summary indicator of the mechanics of human pathological gait. Gait Posture. 2000 Dec;12(3):243-50. doi: 10.1016/s0966-6362(00)00081-3. PMID 11154935
- [Background] Farris DJ, Hampton A, Lewek MD, Sawicki GS. Revisiting the mechanics and energetics of walking in individuals with chronic hemiparesis following stroke: from individual limbs to lower limb joints. J Neuroeng Rehabil. 2015 Feb 27;12:24. doi: 10.1186/s12984-015-0012-x. PMID 25889030
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Frazzitta G, Balbi P, Maestri R, Bertotti G, Boveri N, Pezzoli G. The beneficial role of intensive exercise on Parkinson disease progression. Am J Phys Med Rehabil. 2013 Jun;92(6):523-32. doi: 10.1097/PHM.0b013e31828cd254. PMID 23552330
- [Background] Gallo PM, McIsaac TL, Garber CE. Walking economy during cued versus non-cued self-selected treadmill walking in persons with Parkinson's disease. J Parkinsons Dis. 2014;4(4):705-16. doi: 10.3233/JPD-140445. PMID 25261459
- [Background] Gomenuka NA, Bona RL, da Rosa RG, Peyre-Tartaruga LA. The pendular mechanism does not determine the optimal speed of loaded walking on gradients. Hum Mov Sci. 2016 Jun;47:175-185. doi: 10.1016/j.humov.2016.03.008. Epub 2016 Mar 24. PMID 27017543
- [Background] Hackney ME, Kantorovich S, Levin R, Earhart GM. Effects of tango on functional mobility in Parkinson's disease: a preliminary study. J Neurol Phys Ther. 2007 Dec;31(4):173-9. doi: 10.1097/NPT.0b013e31815ce78b. PMID 18172414
- [Background] Hausdorff JM, Schaafsma JD, Balash Y, Bartels AL, Gurevich T, Giladi N. Impaired regulation of stride variability in Parkinson's disease subjects with freezing of gait. Exp Brain Res. 2003 Mar;149(2):187-94. doi: 10.1007/s00221-002-1354-8. Epub 2003 Jan 22. PMID 12610686
- [Background] Herman T, Giladi N, Gruendlinger L, Hausdorff JM. Six weeks of intensive treadmill training improves gait and quality of life in patients with Parkinson's disease: a pilot study. Arch Phys Med Rehabil. 2007 Sep;88(9):1154-8. doi: 10.1016/j.apmr.2007.05.015. PMID 17826461
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Kuo AD, Donelan JM. Dynamic principles of gait and their clinical implications. Phys Ther. 2010 Feb;90(2):157-74. doi: 10.2522/ptj.20090125. Epub 2009 Dec 18. PMID 20023002
- [Background] Merello M, Fantacone N, Balej J. Kinematic study of whole body center of mass position during gait in Parkinson's disease patients with and without festination. Mov Disord. 2010 Apr 30;25(6):747-54. doi: 10.1002/mds.22958. PMID 20222128
- [Background] MONTEIRO, E.P et al. Aspectos biomecânicos da locomoção de pessoas com doença de Parkinson: revisão narrativa. Revista Brasileira de Ciências do Esporte, ago. 2016. doi.org/10.1016/j.rbce.2016.07.003
- [Background] Monteiro EP, Franzoni LT, Cubillos DM, de Oliveira Fagundes A, Carvalho AR, Oliveira HB, Pantoja PD, Schuch FB, Rieder CR, Martinez FG, Peyre-Tartaruga LA. Effects of Nordic walking training on functional parameters in Parkinson's disease: a randomized controlled clinical trial. Scand J Med Sci Sports. 2017 Mar;27(3):351-358. doi: 10.1111/sms.12652. Epub 2016 Feb 2. PMID 26833853
- [Background] Morris M, Iansek R, McGinley J, Matyas T, Huxham F. Three-dimensional gait biomechanics in Parkinson's disease: evidence for a centrally mediated amplitude regulation disorder. Mov Disord. 2005 Jan;20(1):40-50. doi: 10.1002/mds.20278. PMID 15390033
- [Background] PEYRÉ-TARTARUGA, L.A; MONTEIRO, E.P. PERSPECTIVE: A new integrative approach to evaluate pathological gait: locomotor rehabilitation index. Clinical Trials in Degenerative Diseases, jul. 2016. v. 1, n. 2, p. 86-90.
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Reuter I, Mehnert S, Leone P, Kaps M, Oechsner M, Engelhardt M. Effects of a flexibility and relaxation programme, walking, and nordic walking on Parkinson's disease. J Aging Res. 2011;2011:232473. doi: 10.4061/2011/232473. Epub 2011 Mar 30. PMID 21603199
- [Background] Saibene F, Minetti AE. Biomechanical and physiological aspects of legged locomotion in humans. Eur J Appl Physiol. 2003 Jan;88(4-5):297-316. doi: 10.1007/s00421-002-0654-9. Epub 2002 Nov 13. PMID 12527959
- [Background] SCHEPENS, B. et al. Mechanical work and muscular efficiency in walking children. The Journal of Experimental Biology, fev. 2004. v. 207, n. Pt 4, p. 587-96. SHANAHAN, J. et al. Dance for people with Parkinson disease: What is the evidence telling us? Archives of Physical Medicine and Rehabilitation, jan. 2015 v. 96, p. 141-53.
- [Background] Sharp K, Hewitt J. Dance as an intervention for people with Parkinson's disease: a systematic review and meta-analysis. Neurosci Biobehav Rev. 2014 Nov;47:445-56. doi: 10.1016/j.neubiorev.2014.09.009. Epub 2014 Sep 28. PMID 25268548
- [Background] Shine JM, Moore ST, Bolitho SJ, Morris TR, Dilda V, Naismith SL, Lewis SJ. Assessing the utility of Freezing of Gait Questionnaires in Parkinson's Disease. Parkinsonism Relat Disord. 2012 Jan;18(1):25-9. doi: 10.1016/j.parkreldis.2011.08.002. Epub 2011 Aug 26. PMID 21872523
- [Background] SOARES, G.S.; PEYRÉ-TARTARUGA, L.A. Doença de Parkinson e exercício físico: uma revisão de literatura. Ciência em Movimento, 2010. v. 24, p. 69-86.
- [Background] Tuon T, Valvassori SS, Dal Pont GC, Paganini CS, Pozzi BG, Luciano TF, Souza PS, Quevedo J, Souza CT, Pinho RA. Physical training prevents depressive symptoms and a decrease in brain-derived neurotrophic factor in Parkinson's disease. Brain Res Bull. 2014 Sep;108:106-12. doi: 10.1016/j.brainresbull.2014.09.006. Epub 2014 Sep 28. PMID 25264157
- [Background] Wild LB, de Lima DB, Balardin JB, Rizzi L, Giacobbo BL, Oliveira HB, de Lima Argimon II, Peyre-Tartaruga LA, Rieder CR, Bromberg E. Characterization of cognitive and motor performance during dual-tasking in healthy older adults and patients with Parkinson's disease. J Neurol. 2013 Feb;260(2):580-9. doi: 10.1007/s00415-012-6683-3. Epub 2012 Sep 29. PMID 23052601
- [Background] Willems PA, Cavagna GA, Heglund NC. External, internal and total work in human locomotion. J Exp Biol. 1995 Feb;198(Pt 2):379-93. doi: 10.1242/jeb.198.2.379. PMID 7699313
- [Background] Zigmond MJ, Smeyne RJ. Exercise: is it a neuroprotective and if so, how does it work? Parkinsonism Relat Disord. 2014 Jan;20 Suppl 1:S123-7. doi: 10.1016/S1353-8020(13)70030-0. PMID 24262162
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886